CLINICAL TRIAL: NCT04764721
Title: Characterization in 18F-FDG PET-CT of Brain and Lung Lesions in Young Subjects With Sequelae Psycho-cognitive Disorders in the Aftermath of Severe Covid-19
Brief Title: Characterization in 18F-FDG PET-CT of Brain and Lung Lesions in Subjects With a History of Severe COVID-19
Acronym: TEP-COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A2021-01-01
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Covid-19
Keywords: Covid-19; brain; 18F-FDG PET-CT; lung
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients with sequential psycho-cognitive disorders following severe COVID-19 and included in the Neurocog-Covid study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients enrolled in Neurocog-Covid study in Nancy hospital (Experimental): Young patients (< 65 year old) who contracted VIDOC 19 and were hospitalized for less than 7 days during the first wave, and who present cognitive disorders may be definitively included in the Neurocog-Covid study if their neuropsychological assessment is abnormal. They will then have a prescription for a cerebral MRI and will be enrolled in the TEP-Covid study. If they accept, they will receive a 18F-FDG PET-CT .
  Interventions: Device: 18F-FDG PET-CT

INTERVENTIONS:
Device: 18F-FDG PET-CT — Enrolled patients in Neurocog-Covid will receive a 18F-FDG PET-CT

SUMMARY:
Patients with Covid-19 (Coronavirus disease 19) may experience multiple neurological symptoms .

18F-FDG PET-CT ( Positons EmissionTomography coupled with a Computer Tomography with flurodesoxyglucose labelled with fluor 18), which reflects neuronal glycolytic metabolism, shows early variations in neuronal function.

Moreover the tropism of Covid-19 is essentially pulmonary and the hypothesis of this study is with 18F-FDG PET-CT it's possible to study the relationship between cerebral metabolism and the metabolism of pulmonary lesions following Covid-19 infection.

DETAILED DESCRIPTION:
Patients with Covid-19 may experience multiple neurological symptoms including confusion and headaches (non-specific neurological symptoms), while others develop specific neurological manifestations, including stroke, related to increased bleeding disorders, seizures and signs of encephalitis.

The coronavirus enters the central nervous system through the olfactory bulb, causing olfactory and taste dysfunctions. These symptoms may appear before, during or even after the general symptoms.

Indeed, 18F-FDG PET-CT, which reflects neuronal glycolytic metabolism, shows early variations in neuronal function, even in the absence of morphological changes visualized by MRI (Magnetic Resonance Imaging).

Moreover the tropism of Covid-19 is essentially pulmonary and it is accepted that acute pulmonary lesions are independent risk factors for cerebral hypoxia. Furthermore, the cytokine storm due to COVID-19 and the resulting hyperinflammation state may induce a transient increase in pressure, with endothelial and vascular lesions and increased capillary permeability, and promote pulmonary oedema leading to secondary cerebral damage.

The lung/brain relationship is therefore essential to be studied in pathologies whose main tropism is the lung.

18F-FDG PET has the advantage of being able to explore both cerebral metabolism and the metabolism of COVID-19-related lung lesions.

The hypothesis of this study is that 18F-FDG PET-CT can objectify and characterize central nervous system involvement in Covid-19 infection. It also makes it possible to study the relationship between cerebral metabolism and the metabolism of pulmonary lesions following Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* Patient included in the Neurocog-Covid study (i.e. presenting a cognitive disorder that has been objectified on the neuropsychological assessment and having to undergo a cerebral MRI),
* Patient who has received full information about the organization of the research and has given written informed consent (or a third person, independent of the investigator and sponsor, in the case of literacy disability),
* Patient affiliated to or beneficiary of a social security plan

Exclusion Criteria:

* Women of childbearing age who do not have effective contraception.
* Pregnant woman or nursing mother.
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.
* Persons deprived of liberty by a judicial or administrative decision, persons undergoing psychiatric care pursuant to articles L. 3212-1 and L. 3213-1
* Contraindication to perform 18F-FDG PET-CT
* Patients with a history of pre-Covid-19 psychiatric or chronic illness
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
To characterize the changes in brain metabolism in 18F-FDG PET-CT in patients enrolled in Neurocog-Study in the hospital of Nancy | 13 months
  Volumes and topographies of brain with a decrease in glycolytic metabolism in 18F-FDG PET-CT compared to the brain metabolism of a control population.

SECONDARY OUTCOMES:
To compare the sensitivity of detection of cerebral abnormalities in MRI and 18F-FDG PET-CT in patients included in Neurocog-Covid study at the hospital of Nancy | 13 months
  Number of abnormal MRI and number of abnormal 18F-FDG PET-CT
To correlate the brain functions impacted on the neuropsychological assessment to the brain metabolism in 18F-FDG PET-CT in patients included in the Neurocog-Covid study at the Nancy Hospital | 13 months
  Volumes and topographies of brain with a decrease in glycolytic metabolism in 18F-FDG PET-CT in relation to cognitive profiles identified as deficient.
Correlating brain metabolism to the volume of damage to the lung sequelae of Covid-19. | 13 months
  Volumes and topographies of brain with a decrease in glycolytic metabolism in 18F-FDG PET-CT in relation to the volumes affected in the lungs

CONTACTS AND LOCATIONS:
Overall Officials: Antoine VERGER, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU NANCY Brabois, nuclear medicine department, Vandœuvre-lès-Nancy, France